CLINICAL TRIAL: NCT06101732
Title: Breast Reconstruction by Lipomodeling Alone or With Flap: Evaluation in Franche-Comté
Brief Title: LIMBO : Breast Reconstruction by Lipomodeling Alone or With Flap: Evaluation in Franche-Comté
Acronym: LIMBO
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: 2022/684
Record Dates: First submitted 2023-10-17; First posted 2023-10-26 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-01

CONDITIONS: Breast Cancer; Surgery
Keywords: lipodelling; breast reconstruction
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Limbo study is a retrospective descriptive study which aims to establish the current state of breast reconstruction surgery at the Besançon University Hospital and Hôpital Nord Franche-Comté, between October 2017 and December 2021.

ELIGIBILITY:
Inclusion Criteria:

* Patient who has undergone breast reconstruction using lipomodelling alone or in association with a flap (greater dorsal, DIEP Deep Inferior Epigastric Perforator flap or TRAM Tranverse Rectus Abdominis Myocutaneous Flap), since October 2017.

Patient whose follow-up in plastic surgery is considered completed (final result obtained, patient lost to follow-up or not wishing to continue) at the time of data collection.

Exclusion Criteria:

* Patient under 18 at first consultation
* Opposition of the patient to the collection of her data

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Patient who has undergone breast reconstruction using lipomodelling alone or in association with a flap (greater dorsal, DIEP Deep Inferior Epigastric Perforator flap or TRAM Tranverse Rectus Abdominis Myocutaneous Flap)
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2022-10-13 (Actual); Study Completion 2022-10-13 (Actual)

PRIMARY OUTCOMES:
number of surgical procedures according to the type of breast reconstruction using lipomodelling alone or in combination with a flap | Between october 2017 and 2022
  number of surgical procedures

SECONDARY OUTCOMES:
description of patients' age | at inclusion
  patient age
description of patients' Body Mass Index | at inclusion
  Body Mass Index
description of patients' menopause status | at the time of data collection
  menopause status
description of patients' smoking status | at inclusion
  smoking status
description of patients' diabetes or other medical condition | at inclusion
description of patients' relevant medical history | at inclusion
  relevant medical history
description of patients' History of breast surgery | at inclusion
  hsitory of breast surgery
description of patients' type of cancer | at inclusion
  cancer histology
description of patients' type of surgical treatment | at inclusion
  type of breast reconstruction using lipomodelling alone or in combination with a flap
description of patients' Type of treatment associated with surgery | at inclusion
  Type of treatment associated with surgery
description of Time elapsed between mastectomy and reconstruction | at inclusion
  number of month between the date of mastectomy and date of reconstruction

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de besancon, Besançon, France